CLINICAL TRIAL: NCT07332390
Title: Comparison of Moderate Load Eccentric Core Exercises and Pilates in Patients With Non-Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/26
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate load eccentric core exercises (Experimental): Participants will perform moderate load eccentric core exercises targeting trunk stabilizer and global core muscles, including eccentric back extensions, abdominal rollouts etc. Exercises will emphasize slow eccentric contractions (3-5 sec) at 50-70% 1RM or equivalent resistance, performed for 8-12 reps, 2-3 sets, three times per week. The protocol aims to enhance core strength, proprioception, neuromuscular control, and spinal stability, thereby reducing pain, disability, and recurrence in nonspecific low back pain.
  Interventions: Procedure: MODERATE LOAD ECCENTRIC CORE EXERCISES
- Pilates (Experimental): Participants will undergo a Pilates-based exercise program focusing on core activation, controlled breathing, postural alignment, and trunk stability. The program will include mat-based Pilates movements such as pelvic tilts, bridging, hundred, leg stretch, and spine mobility exercises. Sessions will emphasize slow, controlled movements with deep stabilizer activation (transversus abdominis, multifidus), performed for 8-12 reps, 2-3 sets, three times per week. The aim is to improve core strength, posture, proprioception, flexibility, and overall functional control, leading to reduced pain and disability in nonspecific low back pain.
  Interventions: Procedure: Pilates

INTERVENTIONS:
Procedure: MODERATE LOAD ECCENTRIC CORE EXERCISES — MODERATE LOAD ECCENTRIC CORE EXERCISES: Eccentric training protocol will be incorporated in core strengthening regime . This will be conducted in two phases. Phase 1 will be the familiarization phase and phase 2 will be the acclimatization phase .
  Arms: Moderate load eccentric core exercises
Procedure: Pilates — Pilates description: participants will be enrolled in group B of the study and will follow a Pilates program designed to ensure progressive overload. The protocol will begin with foundational exercises focused on motor learning and core activation, progressing gradually to more advanced functional and load-bearing stability exercises. The primary focus will be on deep core recruitment, utilizing a beginner-level approach to avoid generalized movements and ensure targeted muscle activation. This structured progression will ensure that core stability remains the central focus, with each phase building upon the previous one.
  Warm up:
  Before starting the session, participants will perform warm up exercises for 10 minutes that include the following exercises:
  1. Seated trunk rotation.
  2. Standing trunk rotation
  3. High knees
  4. Standing side bends
  5. Standing back stretch Each exercise will be performed 10 -12 times on each side. Cool down: Child's pose,Cat-cow stretch,Knee to chin
  Arms: Pilates

SUMMARY:
Low back pain (LBP) is a major global health concern, significantly affecting mobility, productivity, and quality of life. Non-specific low back pain (NSLBP), which accounts for most LBP cases, is associated with impaired proprioception, reduced lumbar range of motion (ROM), decreased muscular endurance, and altered neuromuscular control. Joint position error (JPE) is a key indicator of proprioceptive dysfunction, contributing to postural instability and movement impairments in NSLBP patients. Effective rehabilitation strategies are essential to improve functional outcomes and prevent recurrence. Exercise therapy, particularly core stabilization exercises, plays a crucial role in NSLBP management. Among various approaches, moderate-load eccentric core exercises and Pilates have gained attention for their potential benefits. Eccentric exercises improve neuromuscular control, proprioception, and endurance by emphasizing controlled muscle lengthening. Pilates, on the other hand, focuses on core activation, postural alignment, and flexibility to enhance spinal stability and movement efficiency. However, limited research directly compares their effects on joint position error, pain, lumbar ROM, and core endurance in NSLBP patients. This randomized controlled trial (RCT) will recruit 44 NSLBP patients from Fauji Foundation Hospital, Rawalpindi, using purposive sampling. Participants will be randomly assigned to either the moderate-load eccentric core exercise group or the Pilates group for an 8-week supervised intervention. Assessments will be conducted at baseline, the 4th week, and post-intervention using an inclinometer (JPE), NPRS (pain), an inclinometer (lumbar ROM), and McGill Torso Endurance Battery (core endurance). SPSS version 21.0 will be used to analyze the data, with normality assessed through the Shapiro-Wilk test or the Kolmogorov-Smirnov test. Group differences will be analyzed using an Independent Sample t-test for normally distributed data and Mann-Whitney U test in case of non-normally distributed data (p < 0.05).

DETAILED DESCRIPTION:
Low back pain (LBP) is the most prevalent musculoskeletal condition worldwide, affecting an estimated 619 million people and ranking among the leading causes of disability across all ages. It reduces quality of life, productivity, and mental well-being, creating a major socioeconomic burden. The biopsychosocial model describes LBP as a multifactorial disorder influenced by biological, psychological, and social factors, emphasizing the need for interdisciplinary management. According to the WHO, LBP is defined as pain occurring between the 12th rib and inferior gluteal folds, with or without referred pain, and is classified as acute (<6 weeks), subacute (6-12 weeks), or chronic (>12 weeks).

Most LBP is nonspecific (≈90%), with no structural cause, and influenced by inactivity, obesity, smoking, and psychosocial stress. In 2019, LBP ranked 6th in DALYs for females, highlighting a greater burden among women. Impaired trunk muscle activation and proprioception contribute to motor control deficits, abnormal recruitment patterns, and recurrent pain. Core musculature plays a central role: Bergmark classified spinal muscles into deep stabilizers (e.g., multifidus, transversus abdominis) and superficial movers (e.g., extensors), both essential for spinal stability. Weakness of extensors predisposes to initial episodes of LBP, while dysfunction of deep stabilizers is associated with chronicity. Exercise therapy is a key intervention. Eccentric training has gained attention for superior neuromuscular adaptations, increasing strength, muscle fiber size, and coordination, with evidence from athletic populations showing functional benefits beyond concentric training. Pilates provides a holistic approach emphasizing controlled movement, breathing, and core activation, improving alignment, flexibility, proprioception, and quality of life. Core stabilization exercises (CSE) specifically target proprioception and motor control, reducing lumbar joint position error, pain, and disability.

Several randomized controlled trials support these interventions. Puntumetakul et al. reported that CSE significantly reduced lumbar JPE, pain, and disability compared to thermal therapy. Zirek et al. found that six weeks of Pilates decreased pain and disability and improved quality of life in chronic LBP. Su Su Hlaing et al. showed that core stabilization and strengthening improved proprioception and muscular thickness of TrA and multifidi. Antonelli et al. demonstrated that Pilates improved pelvic alignment, trunk stability, and reduced pain. Moradi et al. confirmed that modified Pilates led to greater improvements in motor control, pain, and functional recovery compared to traditional exercises.

ELIGIBILITY:
Inclusion Criteria:

* • Adults 18 to 45 years

  * Both genders
  * Low back (from T12 to buttock line) pain for more than 3 months
  * Non-specific low back pain i.e. signs or symptoms not attributable to any specific structure
  * Low back pain on 3-8 NPRS

Exclusion Criteria:

* • Acute flare Low Back Pain

  * Low back pain on NPRS (>8)
  * Thoracic pain
  * Centralization and peripheralization of pain
  * Leg symptoms when walking, eased in flexion (Signs of stenosis)
  * Pain due to repetitive movement
  * Paresthesia/numbness
  * Structural deformity (scoliosis, spondylosis, spondylolisthesis)
  * Curve reversal
  * Pregnancy
  * Post-surgery (within 6 months of abdominal, spinal, or lower limb surgery)
  * Degenerative or inflammatory spinal diseases
  * Malignancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline , 4th week and 8th week.
  it will be assessed by Numeric Pain Rating Scale NPRS. 0 means no pain and 10 means worst pain.
Lumber range of motion | Baseline , 4th week and 8th week.
  Lumber range of motion will be measured through dual inclinometer. Ranges include lumber flexion, lumber extension, right lateral flexion and left lateral flexion.
Core endurance | baseline , 4th week and 8th week
  It will be assessed through McGill core endurance battery. Core endurance will be assessed by measuring the time to hold a certain position. Time will be recorded.
  Core endurance include:
  Flexor trunk endurance Extensor trunk endurance Right side plank Left side plank
Inclinometer For Lumbar Joint Position Error | BASELINE, 4th and 8th week
  Two inclinometers will be used for measuring JPE, one will be positioned at T12 spinous process and other will be placed at S1 spinous process. Participants will be blindfolded to eliminate visual cues and will memorize a target position by holding it for 5 seconds before returning to neutral. They will then attempt to reposition their spine into the target position in lumber flexion without visual feedback. The difference between the achieved and target positions will be recorded as the joint position error, measuring proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan